CLINICAL TRIAL: NCT00001197
Title: Effect of Hydroxyurea on Fetal Hemoglobin Synthesis in Patients With Sickle Cell Anemia
Brief Title: Hydroxyurea for the Treatment of Patients With Sickle Cell Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 840029; 84-H-0029
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-05-18

CONDITIONS: Sickle Cell Anemia
Keywords: Gene Expression Therapy; Gamma Globin Gene; Hemoglobin Switching; Bone Marrow; Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea

SUMMARY:
A total of fifty severely affected patients with homozygous sickle cell disease or other sickling disorders (e.g. B negative or B positive Thalassemia/Sickle) who are greater than 18 years of age will be eligible for treatment. Such patients must be able to tolerate an extensive period without blood transfusion and have relatively well preserved renal and hepatic function (creatinine less than 1.5 mg/dl and normal liver function test with exception of a mild elevation in transaminase). Evidence of severe sickle cell anemia will include recurrent pain crisis, chronic bone oain, evidence of aseptic necrosis with symptoms, and intractable leg ulcer, etc.

On admission to the study, each patient will receive a complete history and physical examination. These data and standard laboratory evaluation, including a test for pregnancy if appropriate, will be adequate to ascertain whether any of the criteria for exclusion are present. Each patient must accept responsibility for for using an effective means of contraception. Patients who are found to be HIV positive will be excluded from the study....

DETAILED DESCRIPTION:
Hydroxyurea is a cell-cycle specific agent that blocks DNA synthesis by inhibiting ribonucleotide reductase, the enzyme that converts ribonucleotides to deoxyribonucleotides. Hydroxyurea has been shown to induce the production of HbF, initially in non-human primates, and now in more than fifty patients with sickle cell anemia. The majority of patients with sickle cell disease respond to the drug with a more than two-fold increase in HbF levels; in some patients the percent of HbF exceeds 10 or 15 percent. It is estimated that levels of 20 percent are required to substantially reduce the sickling propensity of red cells and to modulate disease severity. We propose now to treat several patients chronically with hydroxyurea to monitor the durability of the response, to examine for unanticipated long term sided effects and to determine hematological changes occurring longitudinally. Such patients will be candidates for protocols determining the ability of other agents to enhance HbF synthesis, especially in hydroxyurea non-responders. Finally, a series of in vitro studies are planned to attempt to develop predictors of response.

ELIGIBILITY:
* INCLUSION CRITERIA:

A total of fifty severely affected patients with homozygous sickle cell disease or other sickling disorders (e.g., B negative or B positive Thalassemia/Sickle) who are greater than 18 years of age will be eligible for treatment. Such patients must be able to tolerate an extensive period without blood transfusion and have relatively well preserved renal and hepatic function (creatinine less than 1.5 mg/dl and normal liver function test with exception of a mild elevation in transaminase). Evidence of severe sickle cell anemia will include recurrent pain crisis, chronic bone pain, evidence of aseptic necrosis with symptoms, and intractable leg ulcers, etc.

EXCLUSION CRITERIA:

Patients who are found to be HIV positive will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1984-02-07; Primary Completion 2003-12-21 (Actual); Study Completion 2015-05-18 (Actual)

PRIMARY OUTCOMES:
An increment in fetal hemoglobin production as a result of hydroxyurea.

CONTACTS AND LOCATIONS:
Overall Officials: Griffin P Rodgers, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rodgers GP, Dover GJ, Noguchi CT, Schechter AN, Nienhuis AW. Hematologic responses of patients with sickle cell disease to treatment with hydroxyurea. N Engl J Med. 1990 Apr 12;322(15):1037-45. doi: 10.1056/NEJM199004123221504. PMID 1690857
- [Background] Fibach E, Burke LP, Schechter AN, Noguchi CT, Rodgers GP. Hydroxyurea increases fetal hemoglobin in cultured erythroid cells derived from normal individuals and patients with sickle cell anemia or beta-thalassemia. Blood. 1993 Mar 15;81(6):1630-5. PMID 7680923
- [Background] Rodgers GP, Dover GJ, Uyesaka N, Noguchi CT, Schechter AN, Nienhuis AW. Augmentation by erythropoietin of the fetal-hemoglobin response to hydroxyurea in sickle cell disease. N Engl J Med. 1993 Jan 14;328(2):73-80. doi: 10.1056/NEJM199301143280201. PMID 7677965